CLINICAL TRIAL: NCT00906685
Title: A Prospective, Randomized, Controlled Study on Intravitreal Bevacizumab (Avastin) for Central Retinal Vein Occlusion (CRVO)
Brief Title: Bevacizumab for Central Retinal Vein Occlusion Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anders Kvanta (Other)
Responsible Party: Sponsor-Investigator, Anders Kvanta, Professor, St. Erik Eye Hospital
Organization: St. Erik Eye Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACRVO
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Central Retinal Vein Occlusion
Keywords: CRVO; anti-VEGF; Macular edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravitreal bevacizumab (Active Comparator)
  Interventions: Drug: bevacizumab
- Sham injection (Sham Comparator)
  Interventions: Drug: Sham bevacizumab injection

INTERVENTIONS:
Drug: bevacizumab — Intravitreal injection of 1.25 mg bevacizumab
  Arms: Intravitreal bevacizumab
Drug: Sham bevacizumab injection — Sham intravitreal injection
  Arms: Sham injection

SUMMARY:
Central retinal vein occlusion is a leading cause of severe visual impairment. Until now, no treatment has been available to improve visual acuity. The present study intends to investigate if intravitreal bevacizumab can improve visual acuity as compared to sham-treated control patients.

ELIGIBILITY:
Inclusion Criteria:

* CRVO with duration < 6 months
* Visual acuity of 20/800 to 20/50

Exclusion Criteria:

* CRVO with duration of > 6 months
* previous treatment with anti-angiogenic drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients gaining 15 ETDRS letters or more | 6 months

SECONDARY OUTCOMES:
Change in foveal thickness | 6 months
Cases of neovascular glaucoma | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kvanta, MD, PhD, Principal Investigator — St Eriks Eye Hospital
Locations (1):
- St Eriks Eye Hospital, Stockholm, Sweden